CLINICAL TRIAL: NCT03028350
Title: A Phase 2 Multicenter, Double-blind, Randomized, Placebo-Controlled Trial to Evaluate Oral Ifetroban in Subjects With Symptomatic Aspirin Exacerbated Respiratory Disease (AERD)
Brief Title: Oral Ifetroban to Treat Aspirin Exacerbated Respiratory Disease (AERD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-IFE-006
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Results first posted 2024-06-28 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Asthma, Aspirin-Induced
MeSH Terms: conditions — Asthma, Aspirin-Induced | interventions — ifetroban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ifetroban Oral Capsule (Experimental): Oral ifetroban, 200 mg daily for 8 weeks
  Interventions: Drug: Ifetroban Oral Capsule
- Placebo Oral Capsule (Placebo Comparator): Oral placebo daily for 8 weeks
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Ifetroban Oral Capsule — Subjects will be treated with oral ifetroban daily for 8 weeks
  Other Names: Ifetroban
  Arms: Ifetroban Oral Capsule
Drug: Placebo Oral Capsule — Subjects will be treated with oral placebo daily for 8 weeks
  Other Names: Placebo
  Arms: Placebo Oral Capsule

SUMMARY:
The purpose of this phase 2 study is to assess the safety and efficacy of oral ifetroban for the treatment of aspirin-exacerbated respiratory disease (AERD). AERD is a disease that involves asthma, recurring nasal polyps, and respiratory reactions to aspirin and other nonsteroidal anti-inflammatory drugs.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind phase 2 trial evaluating approximately 76 subjects with symptomatic AERD on the safety and efficacy of 8 weeks of oral ifetroban treatment. Eligible AERD subjects will be randomized to receive 8 weeks of either oral ifetroban daily or matching placebo followed by a 2-week post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. History of physician-diagnosed asthma
2. History of nasal polyposis
3. History of at least two reactions to oral aspirin or other nonselective cyclooxygenase inhibitor with features of lower airway involvement (cough, chest tightness, wheezing, dyspnea), or one reaction that was life-threatening and required hospitalization, or a diagnosis of AERD by a physician-conducted challenge to aspirin in the last five years before starting treatment.
4. Stable asthma (post-bronchodilator forced expiratory volume in 1 second (FEV1) of ≥ 60%, no glucocorticoid burst for at least two weeks prior to starting treatment, no hospitalizations or emergency room visits for asthma at least three months prior to starting treatment and not on a dose >1000 µg fluticasone or equivalent daily).
5. ≥ 18 years of age
6. Exhibit symptomatic AERD within three weeks of starting treatment by demonstrating a score of at least 20 on the Sino-nasal Outcome Test (SNOT) - 22.

Exclusion Criteria:

1. Current smoking, defined as daily tobacco smoking in the last six months and at least one instance of tobacco smoking in the last three months.
2. Current pregnancy or breastfeeding
3. Use of oral or systemic steroids (e.g. prednisone or equivalent) > 20 mg daily in the last four weeks before starting treatment.
4. Daily use of long-acting antihistamines in the last two weeks before starting treatment.
5. Less than 12 months of allergy shots (maintenance dose of allergy shots are allowed if treatment duration exceeds 12 months). Less than 1 month of 5-lipoxygenase inhibitors (e.g. zileuton) and/or leukotriene receptor antagonists (e.g. montelukast).
6. Any use of nonsteroidal anti-inflammatory drugs (NSAIDs) or any drug that inhibits the cyclooxygenase enzyme in the last two weeks before starting treatment.
7. History of bleeding diathesis or use of anticoagulant or antiplatelet drugs in the last two weeks before starting treatment.
8. Any immunosuppressive treatment including but not limited to methotrexate, cyclosporine, mycophenolate, tacrolimus, gold, penicillamine, sulfasalazine, hydroxychloroquine, azathioprine, and cyclophosphamide in the last two weeks before starting treatment (maintenance dose of allergy shots are allowed if treatment duration exceeds 12 months). Biologics/immunotherapies such as Xolair or Nucala are permitted if duration exceeds three months.
9. Endoscopic sinus surgery / polypectomy within the past three months
10. Previously treated in a clinical trial with ifetroban within the past three months.
11. Previously treated with other investigational drugs within eight weeks or five half-lives, whichever is longer, before screening
12. Conditions/concomitant disease which make them unevaluable for the efficacy endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew White, MD, Principal Investigator — Scripps Research Institute
Locations (16):
- United States (16):
  - Banner University of Arizona Medical Center, Asthma & Airway Disease Research Center, Tucson, Arizona
  - Antelope Valley Clinical Trials, Lancaster, California
  - Scripps Clinic - Carmel Valley, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - The Research Center, Hialeah, Florida
  - Emory University School of Medicine, Sinus, Nasal, and Allergy Center, Atlanta, Georgia
  - Deaconess Clinic, Evansville, Indiana
  - Kansas City Allergy and Asthma Associates, PA, Overland Park, Kansas
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Rochester Regional Health, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ifetroban Oral Capsule | Placebo Oral Capsule
Started | 25 | 29
Completed | 21 | 28
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ifetroban Oral Capsule | Placebo Oral Capsule | Total
Number analyzed (Participants) | 25 | 29 | 54
Age, Continuous [Median (Full Range); unit: years] | 55 [27 to 70] | 45 [24 to 80] | 51 [24 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 11 | 9 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 20 | 25 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 19 | 22 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 29 | 54
Weight [Median (Full Range); unit: kg] | 84.2 [48.2 to 127.3] | 85.4 [52.9 to 137.2] | 84.4 [48.2 to 137.2]
BMI (kg/m2), Categorical >=30; <30 [Count of Participants; unit: Participants]
  >=30 | 11 | 10 | 21
  <30 | 14 | 19 | 33
BMI (kg/m2), Continuous [Median (Full Range); unit: kg/m^2] | 28.8 [18.8 to 43.5] | 27.0 [19.7 to 44.5] | 27.8 [18.8 to 44.5]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sinonasal Outcome Test-22 Score
Description: Sinonasal Outcome Test-22 (SNOT-22) score is a scale with a minimum score of 0 and a maximum score of 110 based on the presence and severity of symptoms and outcomes of rhinosinusitis. Higher scores indicate worse symptoms and/or outcomes.
Time Frame: Baseline and 8 weeks
Population: All subjects enrolled with SNOT-22 measurements at both baseline and 8 weeks were included. Three enrolled subjects treated with ifetroban did not have SNOT-22 measurements for both timepoints and therefore were not analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ifetroban Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 22 | 29
units on a scale | -6.7 (12.9) | -13.7 (22.6)

2. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire -7 Score
Description: The Asthma Control Questionnaire-7 is a scoring system with a minimum score of 0 and a maximum score of 6 based on the severity and frequency of asthma symptoms. Higher scores indicate worse control of asthma symptoms.
Time Frame: Baseline and 8 weeks
Population: All subjects enrolled with Asthma Control Questionnaire-7 measurements at both baseline and 8 weeks were included. Ten enrolled subjects treated with ifetroban and 5 enrolled subjects treated with placebo did not have Asthma Control Questionnaire-7 measurements for both timepoints and therefore were not analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ifetroban Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 15 | 24
units on a scale | 0.30 (1.44) | -0.20 (1.01)

3. Secondary Outcome: Change From Baseline in Total Nasal Symptom Score (Morning)
Description: The Total Nasal Symptom Score is a scoring system with a minimum score of 0 and maximum score of 15 based on severity of nasal symptoms. Higher scores indicate worse nasal symptoms.
Time Frame: Baseline and 8 weeks
Population: All subjects enrolled with Total Nasal Symptom Score (morning) measurements at both baseline and 8 weeks were included. Five enrolled subjects treated with ifetroban and 9 enrolled subjects treated with placebo did not have Total Nasal Symptom Score (morning) measurements for both timepoints and therefore were not analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ifetroban Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 20 | 20
units on a scale | -1.28 (1.85) | -2.57 (3.05)

4. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: Change From Baseline in Forced Expiratory Volume in 1 second (FEV1) at 8 weeks
Time Frame: Baseline and 8 weeks
Population: All subjects enrolled with FEV1 measurements at both baseline and 8 weeks were included. Four enrolled subjects treated with ifetroban and 1 enrolled subject treated with placebo did not have FEV1 measurements at both times and therefore were not analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Ifetroban Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 21 | 28
liters | 0.010 (0.421) | 0.004 (0.323)

5. Secondary Outcome: Change From Baseline in Peak Nasal Inspiratory Flow Rate (PNIFR)
Description: Change From Baseline in Peak Nasal Inspiratory Flow Rate (PNIFR) at 8 weeks
Time Frame: Baseline and 8 weeks
Population: All subjects enrolled with PNIFR measurements at both baseline and 8 weeks were included. Five enrolled subjects treated with ifetroban and 1 enrolled subject treated with placebo did not have PNIFR measurements for both timepoints and therefore were not analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | Ifetroban Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 20 | 28
liters/minute | 11.4 (48.3) | -3.70 (29.0)

6. Secondary Outcome: Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO)
Description: Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) at 8 weeks
Time Frame: Baseline and 8 weeks
Population: All subjects enrolled with FeNO measurements at both baseline and 8 weeks were included. Six enrolled subjects treated with ifetroban and 2 enrolled subjects treated with placebo did not have FeNO measurements for both timepoints and therefore were not analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: parts per billion
Arm/Group | Ifetroban Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 19 | 27
parts per billion | 5.70 (9.32) | 1.40 (17.3)

7. Secondary Outcome: Change From Baseline in Total Nasal Symptom Score (Afternoon/Evening)
Description: The Total Nasal Symptom Score is a scale with a minimum score of 0 and maximum score of 15 based on severity of nasal symptoms. Higher scores indicate worse nasal symptoms.
Time Frame: Baseline and 8 weeks
Population: All subjects enrolled with Total Nasal Symptom Score (afternoon/evening) measurements at both baseline and 8 weeks were included. Eleven enrolled subjects treated with ifetroban and 6 enrolled subjects treated with placebo did not have Total Nasal Symptom Score (afternoon/evening) measurements for both timepoints and therefore were not analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ifetroban Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 14 | 23
units on a scale | -0.519 (2.28) | -1.58 (2.60)

8. Other Pre Specified Outcome: Change From Baseline in Blood Eosinophil Count
Description: Change From Baseline in Blood Eosinophil Count at 8 Weeks
Time Frame: Baseline and 8 weeks
Population: All subjects enrolled with blood eosinophil measurements at both baseline and 8 weeks were included. Eleven enrolled subjects treated with ifetroban and 13 enrolled subjects treated with placebo did not have blood eosinophil measurements for both timepoints and therefore were not analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: x10^9 cells/liter
Arm/Group | Ifetroban Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 14 | 16
x10^9 cells/liter | 0.00 (0.22) | -0.09 (0.26)

ADVERSE EVENTS:
Time Frame: Through 10 weeks (8 weeks of treatment, 2 weeks of follow-up)
Description: The severity of each event is reported by the investigator according to the following definitions:
  * Mild: Transient symptoms, no interference with the subject's daily activities.
  * Moderate: Marked symptoms, moderate interference with the subject's daily activities.
  * Severe: Considerable interference with the subject's daily activities, unacceptable.
Arm/Group | Ifetroban Oral Capsule | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/29
Other Adverse Events (participants affected / at risk) | 7/25 | 11/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ifetroban Oral Capsule (N=25) | Placebo Oral Capsule (N=29)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ifetroban Oral Capsule (N=25) | Placebo Oral Capsule (N=29)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 4 (5) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (6) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (6)

LIMITATIONS AND CAVEATS:
Planned enrollment for the study was 76 subjects with 38 subjects per treatment arm. Due to enrollment challenges during and following the COVID-19 pandemic, the study was closed with 56 subjects enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT03028350/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT03028350/SAP_001.pdf